CLINICAL TRIAL: NCT05345574
Title: The Effect of Dexmedetomidine and Remifentanil Infusion on Postoperative Sore Throat After Lumbar Spine Surgery in the Prone Position
Brief Title: A Postoperative Sore Throat After Lumbar Spine Surgery in the Prone Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Eun Kyung Choi, Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YUMC 2018-09-029
Record Dates: First submitted 2022-04-19; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Post Operative Sore Throat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine infusion group (Active Comparator): dexmedetomidine infusion (loading dose of 1 ㎍/kg over 10 min and continuous infusion of 0.3-0.6 ㎍/kg/h) during the surgery
  Interventions: Drug: dexmedetomidine infusion
- remifentanil infusion group (Active Comparator): remifentanil of 0.05 ㎍/kg/h during induction, followed by remifentanil infusion (0.05-0.3 ㎍/kg/h) during the surgery
  Interventions: Drug: remifentanil infusion

INTERVENTIONS:
Drug: dexmedetomidine infusion — dexmedetomidine as anaesthetic adjuvant
  Arms: dexmedetomidine infusion group
Drug: remifentanil infusion — remifentanil as anaesthetic adjuvant
  Arms: remifentanil infusion group

SUMMARY:
This study was performed to compare the effect of dexmedetomidine and remifentanil on the incidence and severity of postoperative sore throat in patients undergoing spinal surgery in the prone position who are at risk of developing postoperative sore throat.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status classification I and II
2. Undergoing lumbar spine surgery in prone position

Exclusion Criteria:

1. Pre-existing sore throat, hoarseness, or upper respiratory tract infection
2. Allergy to the study drugs
3. Anticipated difficult airways
4. More than two attempts at intubation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2018-12-26 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative sore throat at rest | 1 hour after surgery
  0=none; 1=occur
incidence of postoperative sore throat at swallowing | 1 hour after surgery
  0=none; 1=occur
severity of postoperative sore throat at rest | 1 hour after surgery
  4-point scale (0=none; 1=mild; 2=moderate; 3=severe)
severity of postoperative sore throat at swallowing | 1 hour after surgery
  4-point scale (0=none; 1=mild; 2=moderate; 3=severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Eun kyung Choi, Daegu, Korea (the Republic Of), South Korea